CLINICAL TRIAL: NCT02339233
Title: Spinal Epidural Electrode Array to Facilitate Standing and Stepping After Spinal Cord Injury
Brief Title: Epi Stim to Facilitate Standing and Stepping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: University of California, Los Angeles (Other); Christopher Reeve Paralysis Foundation (Other); Kessler Foundation (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Susan Harkema, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07.0066 Epi Stim; 5R01EB007615 (NIH)
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Results first posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Spinal Cord Injury
Keywords: Epidural Stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epidural Stimulator (Experimental): Eligible participants will be implanted with 16-electrode epidural array in the T11-L1 area of the spinal cord
  Interventions: Device: Standing and Stepping with spinal cord Epidural Stimulation

INTERVENTIONS:
Device: Standing and Stepping with spinal cord Epidural Stimulation — Standing and Stepping with support from trainers as needed, overground or in a harness with body weight support on a treadmill. Epidural stimulation with specific configurations will be administered to generate standing and stepping.
  Other Names: Stand-scES; Step-scES; Locomotor Training (LT)

SUMMARY:
The overall aim is to assess whether task specific locomotor training and spinal cord electrical stimulation (SCES) can induce neural reorganization of the functionally isolated human spinal cord to improve standing and stepping in individuals with functionally complete SCI. The investigators propose that locomotor training will result in generation of more effective standing and stepping efferent patterns by restoring phase dependent modulation of reflexes and reciprocal inhibition, reducing clonus and mediating interlimb coordination. The investigators propose that the SCES will optimize the physiological state of the spinal cord interneuronal circuitry compromised by compensating for loss of supraspinal input for the retraining of these tasks.

DETAILED DESCRIPTION:
Participants will be screened for eligibility and then participate in pre-training motor, bladder and cardiovascular experiments, followed by 80 sessions of locomotor training. Participants will repeat experiments after the 80 training sessions to quantify that no motor pattern changes are achievable with locomotor training alone and will be evaluated for appropriate candidacy for surgery and epidural stimulation. Participants will be surgically implanted with an epidural stimulator and experiments will be conducted with and without stimulation. Investigators will identify appropriate stimulation parameters for inducing stepping and standing in combination with manual assistance using body weight support on a treadmill and/or overground. Participants will undergo 80-200 training sessions of locomotor training with epidural stimulation. Experiments will be repeated mid and post-training interventions.

ELIGIBILITY:
Inclusion Criteria:

* All research participants, irrespective of age or sex, will meet the following criteria:

  * stable medical condition without cardiopulmonary disease or dysautonomia that would contraindicate standing or stepping with BWST;
  * no painful musculoskeletal dysfunction, unhealed fracture, contracture, pressure sore, or urinary tract infection that might interfere with stand or step training;
  * no clinically significant depression or ongoing drug abuse;
  * no current anti-spasticity medication regimen;
  * non-progressive SCI above T10;
  * must not have received botox injections in the prior six months;
  * be unable to stand or step independently;
  * at least one-year post injury; and
  * must be at least 18 years of age.

In addition, all subjects must satisfy each of the three conditions of the functional neurophysiological assessment described below.

Functional Neurophysiological Assessment (FNPA). We will use FNPA to screen potential research participants based on specific neurophysiological inclusion criteria. Participants must have no volitional control of movement below the level of the lesion, but must retain some brain influence on spinal reflexes. Our target population, which will be identified by FNPA, cannot be identified reliable using traditional assessments: hence individual subjects may be classified widely as Class A, B, or C on the ASIA SCI scale. We will include only subjects who fulfill the following three requirements:

* There is no descending volitional control of movement below the lesion
* Segmental reflexes remain functional below the lesion
* Brain influence on spinal reflexes is retained

Exclusion Criteria:

* Ventilatory dependent
* painful musculoskeletal function, unhealed fracture, contracture, or pressure sore that might interfere with training;
* clinically significant depression or ongoing drug abuse;
* cardiovascular, respiratory, bladder or renal disease unrelated to SCI;
* severe anemia (Hgb<8 g/dL) or hypovolemia; and
* HIV or AIDS related illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Harkema, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Background] Herrity AN, Williams CS, Angeli CA, Harkema SJ, Hubscher CH. Lumbosacral spinal cord epidural stimulation improves voiding function after human spinal cord injury. Sci Rep. 2018 Jun 6;8(1):8688. doi: 10.1038/s41598-018-26602-2. PMID 29875362
- [Background] Mesbah S, Angeli CA, Keynton RS, El-Baz A, Harkema SJ. A novel approach for automatic visualization and activation detection of evoked potentials induced by epidural spinal cord stimulation in individuals with spinal cord injury. PLoS One. 2017 Oct 11;12(10):e0185582. doi: 10.1371/journal.pone.0185582. eCollection 2017. PMID 29020054
- [Background] Sayenko DG, Angeli C, Harkema SJ, Edgerton VR, Gerasimenko YP. Neuromodulation of evoked muscle potentials induced by epidural spinal-cord stimulation in paralyzed individuals. J Neurophysiol. 2014 Mar;111(5):1088-99. doi: 10.1152/jn.00489.2013. Epub 2013 Dec 11. PMID 24335213
- [Result] Angeli CA, Edgerton VR, Gerasimenko YP, Harkema SJ. Altering spinal cord excitability enables voluntary movements after chronic complete paralysis in humans. Brain. 2014 May;137(Pt 5):1394-409. doi: 10.1093/brain/awu038. Epub 2014 Apr 8. PMID 24713270
- [Result] Angeli CA, Boakye M, Morton RA, Vogt J, Benton K, Chen Y, Ferreira CK, Harkema SJ. Recovery of Over-Ground Walking after Chronic Motor Complete Spinal Cord Injury. N Engl J Med. 2018 Sep 27;379(13):1244-1250. doi: 10.1056/NEJMoa1803588. Epub 2018 Sep 24. PMID 30247091
- [Result] Rejc E, Angeli CA, Atkinson D, Harkema SJ. Motor recovery after activity-based training with spinal cord epidural stimulation in a chronic motor complete paraplegic. Sci Rep. 2017 Oct 26;7(1):13476. doi: 10.1038/s41598-017-14003-w. PMID 29074997
- [Result] Rejc E, Angeli CA, Bryant N, Harkema SJ. Effects of Stand and Step Training with Epidural Stimulation on Motor Function for Standing in Chronic Complete Paraplegics. J Neurotrauma. 2017 May 1;34(9):1787-1802. doi: 10.1089/neu.2016.4516. Epub 2016 Oct 5. PMID 27566051
- [Result] Rejc E, Angeli C, Harkema S. Effects of Lumbosacral Spinal Cord Epidural Stimulation for Standing after Chronic Complete Paralysis in Humans. PLoS One. 2015 Jul 24;10(7):e0133998. doi: 10.1371/journal.pone.0133998. eCollection 2015. PMID 26207623
- [Result] Harkema S, Gerasimenko Y, Hodes J, Burdick J, Angeli C, Chen Y, Ferreira C, Willhite A, Rejc E, Grossman RG, Edgerton VR. Effect of epidural stimulation of the lumbosacral spinal cord on voluntary movement, standing, and assisted stepping after motor complete paraplegia: a case study. Lancet. 2011 Jun 4;377(9781):1938-47. doi: 10.1016/S0140-6736(11)60547-3. Epub 2011 May 19. PMID 21601270

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Epidural Stimulator
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Epidural Stimulator
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Lower Extremity Independence Time During 10 Min Standing Bout After 160 Sessions (1 Year)
Description: We will measure the amount of time individuals are able to stand without manual assistance (independently) throughout a 10 min bout
Time Frame: Baseline, 160 sessions (1 year)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Epidural Stimulator
Number analyzed (Participants) | 8
minutes | 40.6 (30.2)

2. Primary Outcome: Change From Baseline of Stepping Independence Time During 6 Min Stepping Bout After 160 Sessions (1 Year)
Description: We will measure the number of steps individuals are able to take without manual assistance (independently) throughout a 6 min stepping bout
Time Frame: Baseline, 160 session (1 year)
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Epidural Stimulator
Number analyzed (Participants) | 8
steps | 197.13 (421.89)

3. Secondary Outcome: Change From Baseline of Number of Consecutive Hip Flexion Repetitions Performed Within One Minute After 160 Sessions (1 Year)
Description: We will measure the ability of the individuals to perform consecutive hip flexion repetitions with stimulation during a 1 minute period
Time Frame: Baseline, 160 sessions (1 year)
Measure: Mean (Standard Deviation); unit: Repetitions
Arm/Group | Epidural Stimulator
Number analyzed (Participants) | 8
Repetitions | 14.25 (9.8)

ADVERSE EVENTS:
Time Frame: From implant through the end of the second intervention, an average of one year.
Arm/Group | Epidural Stimulator
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural Stimulator (N=8)
Device Malfunction (Surgical and medical procedures) | 1 (1)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural Stimulator (N=8)
Muscle Strain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flipped Stimulator (Surgical and medical procedures) | 1 (1)
Electrode Malfunction (Surgical and medical procedures) | 1 (1)
Incision Site Drainage (Skin and subcutaneous tissue disorders) | 1 (1)
Right Ankle Edema (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT02339233/Prot_ICF_000.pdf